CLINICAL TRIAL: NCT01837927
Title: A 52-week Treatment, Multi-center, Randomized, Open Label, Parallel Group Study to Assess the Efficacy of NVA237 (50 μg o.d.) Using Tiotropium (5 μg o.d.) as an Active Control in Brazilian Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease.
Brief Title: Efficacy of NVA237 (50 μg o.d) Using Tiotropium (5μg μg o.d) as Active Control in COPD Patients.
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNVA237ABR01
Record Dates: First submitted 2013-04-18; First posted 2013-04-23 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Efficacy, NVA237, Tiotropium, Chronic Obstructive Pulmonary Disease, COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate; tiotropium-olodaterol

ARMS (2):
- NVA237 (Experimental): NVA237 inhaled via the Breezhaler® device once daily
  Interventions: Drug: NVA237
- Tiotropium (Active Comparator): Tiotropium 5μg inhaled via the Respimat® device once daily
  Interventions: Drug: Tiotropium Respimat®

INTERVENTIONS:
Drug: NVA237 — Once daily for 52 weeks
  Arms: NVA237
Drug: Tiotropium Respimat® — Once daily for 52 weeks
  Arms: Tiotropium

SUMMARY:
This study will assess the Efficacy of NVA237 (50 μg o.d) using tiotropium (5μg μg o.d) as active control in COPD patients.

DETAILED DESCRIPTION:
A 52-week treatment, multicenter, randomized, open-label, parallel-group study to assess the efficacy of NVA237 (50μg once daily) using Tiotropium (5μg once daily) as an active control in Brazilian patients with moderate to severe Chronic Obstructive Pulmonary Disease.

ELIGIBILITY:
Inclusion:

* Men and women aged 40 years or over.
* History of current or former smoking of at least 10 pack-years
* Cooperative outpatients, with a COPD diagnosis established by the measurement of FEV1/FVC < 0.7 post-bronchodilation in basal spirometry (without use of medication or post-washout). Moderate to severe stage patients will be included, with post-bronchodilator FEV1 between 30 and 80% of the normal value according to GOLD 2011 since the inclusion criteria in this trial will be based on spirometry results.

Exclusion:

* Pregnant women or nursing mothers
* History of asthma at visit 1 indicated by, but not limited to:

  * Onset of respiratory symptoms suggestive of asthma (such as coughing, wheezing, shortness of breath) before the age of 40.
  * History of diagnosed asthma
* History of respiratory tract infection within six weeks prior to Visit 1.
* History of hospitalization or emergency care for a COPD exacerbation in the 3 months prior to Visit 1.
* Subjects who require use of home oxygen therapy.
* Patients in the active phase of an assisted pulmonary rehabilitation program and patients who completed the rehabilitation program within 18 months from Visit 1 or 2 of the protocol.17,20
* Patients with known history and diagnosis of alpha-1 antitrypsin deficiency.
* Patients with concomitant lung disease, e.g.: tuberculosis (unless confirmed by radiography as inactive) or clinically significant bronchiectasis.
* Patients who in the investigator's judgment have an abnormality or significant medical condition such as: unstable ischemic heart disease, left ventricular failure, history of myocardial infarction, arrhythmia (except chronic stable atrial fibrillation), history of malignancy of any system (including lung cancer) treated or not within the last 5 years, glaucoma, prostatic hyperplasia, moderate to severe renal impairment, urinary retention, any other condition that might compromise patient safety or compliance, interfere with the evaluations, or prevent the termination of their participation in the study.
* Patients with contraindications to tiotropium or ipratropium treatment or who have experienced undesirable reactions with inhaled anticholinergic agents or patients with a history of an undesirable reaction with sympathomimetic amines or inhaled medication with any of those components, or a history of hypersensitivity to any of the study medications, including rescue medication, or similar classes of medication.
* Patients using tiotropium, long-acting anticholinergics, short-acting anticholinergics, fixed combinations of inhaled beta agonists and inhaled corticosteroids, theophylline. In these cases, the patient is allowed, after agreeing to participate in the study, to enter a washout period from Visit
* Patients using inhaled steroids, alone or as an exchange in a fixed combination at equivalent doses, unless on a stable treatment for at least 1 month prior to randomization
* Patients using nonselective beta-blockers.
* Patients using cromoglycate, nedocromil, ketotifen and leukotriene antagonists unless on stable treatment for at least 1 month prior to randomization .
* Patients who used oral prednisone (or equivalent) over a long period, defined as ≥ 10 mg/day for at least 1 month prior to Visit 1
* Patients who used intramuscular depot corticosteroids within 30 days from Visit 1.
* Patients with a history of long QT Syndrome or with prolonged QTc (> 450 ms) measured at Visit 1 (Fridericia Method).
* Patients who, in the opinion of the investigator, have clinically significant abnormalities on ECG. These patients should not be re-screened.
* Other exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) | Baseline and 12 weeks after treatment.
  Forced expiratory volume in 1 second (FEV1) is the amount of air that can be exhaled in one second. FEV1 will be measured by spirometry. A positive change from baseline in FEV1 indicates improvement in lung function.

SECONDARY OUTCOMES:
Forced Expiratory Volume in 1 Second (FEV1) at day 1 | 30 and 60 minutes post-dose on the first day of study treatment.
  Forced expiratory volume in 1 second (FEV1) is the amount of air that can be exhaled in one second. FEV1 will be measured by spirometry. A positive change from baseline in FEV1 indicates improvement in lung function.
Forced Expiratory Volume in 1 Second (FEV1) at day 7 and weeks 12, 24 and 52 | 30 and 60 minutes post-dose on the 7th day of study treatment and at weeks 12, 24 and 52
  Forced expiratory volume in 1 second (FEV1) is the amount of air that can be exhaled in one second. FEV1 will be measured by spirometry. A positive change from baseline in FEV1 indicates improvement in lung function.
Forced Expiratory Volume in 1 Second (FEV1) at weeks 24 and 52 | pre-dose at weeks 24 and 52 of study treatment
  Forced expiratory volume in 1 second (FEV1) is the amount of air that can be exhaled in one second. FEV1 will be measured by spirometry. A positive change from baseline in FEV1 indicates improvement in lung function.
Change From Baseline in Forced Vital Capacity (FVC) | Days 1 and 7, weeks 12, 24 and 52 of study treatment
  Forced Vital Capacity (FVC) is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. FVC was assessed via spirometry. A positive change from baseline in FVC indicates improvement in lung function.
FEV1 AUC 0-4h | 05, 30, 60 minutes and 4 hours post-dose at days 1, 7 and week 12
  Forced Vital Capacity (FVC) is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. FVC was assessed via spirometry. A positive change from baseline in FVC indicates improvement in lung function.
Safety and tolerance of NVA237 | 52 weeks
  All AEs and SAEs will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals